CLINICAL TRIAL: NCT03346538
Title: Dose Finding Study of MCI-186 in Acute Ischemic Stroke
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business objectives have changed.
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCI-186-J20
Record Dates: First submitted 2017-11-02; First posted 2017-11-17 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Edaravone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Continuous infusion high-dose group (Group H) (Experimental): High-dose MCI-186 will be administered as a bolus, and then as a continuous infusion. In addition, a placebo will be administered as an intravenous infusion twice a day over 30 minutes.
  Interventions: Drug: Continuous infusion high-dose MCI-186; Drug: Approved dosing regimen placebo
- Continuous infusion low-dose group (Group L) (Experimental): Low-dose MCI-186 will be administered as a bolus, and then as a continuous infusion. In addition, a placebo will be administered as an intravenous infusion twice a day over 30 minutes.
  Interventions: Drug: Continuous infusion low-dose MCI-186; Drug: Approved dosing regimen placebo
- Approved dosing regimen group (control group) (Experimental): A placebo will be administered as a bolus, and then as a continuous infusion. In addition, MCI-186 30 mg will be administered as an intravenous infusion twice a day over 30 minutes.
  Interventions: Drug: Continuous infusion placebo; Drug: Approved dosing regimen MCI-186

INTERVENTIONS:
Drug: Continuous infusion high-dose MCI-186 — intravenous injection
  Arms: Continuous infusion high-dose group (Group H)
Drug: Continuous infusion low-dose MCI-186 — intravenous injection
  Arms: Continuous infusion low-dose group (Group L)
Drug: Continuous infusion placebo — intravenous injection
  Arms: Approved dosing regimen group (control group)
Drug: Approved dosing regimen MCI-186 — intravenous injection
  Arms: Approved dosing regimen group (control group)
Drug: Approved dosing regimen placebo — intravenous injection
  Arms: Continuous infusion high-dose group (Group H); Continuous infusion low-dose group (Group L)

SUMMARY:
To investigate the efficacy and safety of MCI-186 (bolus followed by continuous infusion) in acute ischemic stroke patients through a double-blind, parallel-group comparison with the existing MCI-186 dosing regimen (administration twice daily for 14 days) as the control.

ELIGIBILITY:
Inclusion Criteria:

* Patients from whom written consent to study participation has been obtained, either from the patient personally or from the patient's legal guardian
* Patients with age at consent between 20 and 85 years, inclusive
* Patients for whom study treatment can be initiated within 24 hours after onset
* Patients with confirmed new ischemic area only in the supratentorial region on MRI
* Patients with neurological signs equivalent to between 4 and 22, inclusive, on the NIHSS

Exclusion Criteria:

* Patients with disability equivalent to an mRS score of 2 or more from before onset
* Patients being treated with antibiotics for an infection at registration
* Patients who have received or are planning to receive treatment for their primary disease with a prohibited concomitant medication (e.g., a thrombolytic drug) or with a prohibited concomitant therapy (e.g., intravascular therapy)
* Patients for whom the (sub)investigator judges the efficacy endpoints (e.g., NIHSS, mRS, BI) that have been selected for this study can not be measured appropriately, such as patients who are not expected to achieve improvement of 4 or more on the NIHSS because of nerve symptoms that have been present since before the onset of cerebral infarction, Alzheimer's dementia patients, or Parkinson's disease patients
* Patients with severe consciousness disturbances (Japan coma scale ≥ 100)
* Patients with clear concurrent peripheral vascular disease or peripheral neuropathy for whom the (sub)investigator judges the neurological tests could not be performed properly
* Patients with severe renal impairment (e.g., patients with eGFR < 30)
* Patients with severe hepatic impairment (e.g., ALT, AST, or gamma-GTP > 2.5 X ULN)
* Patients with platelet count < 100,000/mm3
* Patients diagnosed by MRI on admission with a disease other than stroke (e.g., intracranial bleeding, subarachnoid bleeding, arteriovenous malformations, Moyamoya disease, brain tumor) or with cerebral aneurysm with a maximum diameter > 7 mm
* Patients with prior or current drug abuse or alcohol dependence
* Patients with prior (or current) malignant tumor within 5 years before stroke onset
* Patients with a past history of hypersensitivity to edaravone drug products
* Patients with concurrent heart disease severe enough to warrant admission and treatment (e.g., acute myocardial infarction, cardiac failure) and with problems with their overall condition judged by the (sub)investigator to be unsuitable for study participation
* Patients for whom MRI tests cannot be performed
* Male or female patients who do not consent to practice contraception from the date of consent until the day after the administration of the last dose of study drug
* Patients who are pregnant or nursing, or who could be pregnant
* Patients who have received other investigational drugs in the 12 weeks prior to consent acquisition
* Patients with body weight ≥ 100 kg
* Patients otherwise judged unsuitable for study participation by the (sub)investigator

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2018-05-14 (Actual); Study Completion 2018-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (45):
- Japan (45):
  - Investigational site 13, Aichi
  - Investigational site 39, Aomori
  - Investigational site 19, Chiba
  - Investigational site 28, Chiba
  - Investigational site 33, Ehime
  - Investigational site 10, Fukui
  - Investigational site 05, Fukuoka
  - Investigational site 09, Fukuoka
  - Investigational site 11, Fukuoka
  - Investigational site 12, Fukuoka
  - Investigational site 18, Fukuoka
  - Investigational site 21, Fukuoka
  - Investigational site 32, Fukuoka
  - Investigational site 37, Fukuoka
  - Investigational site 07, Fukushima
  - Investigational site 08, Fukushima
  - Investigational site 15, Gifu
  - Investigational site 23, Gifu
  - Investigational site 02, Gunma
  - Investigational site 01, Hokkaido
  - Investigational site 22, Hokkaido
  - Investigational site 06, Hyōgo
  - Investigational site 30, Hyōgo
  - Investigational site 42, Hyōgo
  - Investigational site 43, Ishikawa
  - Investigational site 40, Kanagawa
  - Investigational site 24, Kochi
  - Investigational site 35, Miyagi
  - Investigational site 16, Nagano
  - Investigational site 20, Nagano
  - Investigational site 27, Numakunai
  - Investigational site 44, Okayama
  - Investigational site 41, Okinawa
  - Investigational site 03, Osaka
  - Investigational site 25, Osaka
  - Investigational site 38, Saga
  - Investigational site 31, Saitama
  - Investigational site 14, Shimane
  - Investigational site 29, Tochigi
  - Investigational site 36, Tochigi
  - Investigational site 17, Tokyo
  - Investigational site 45, Tokyo
  - Investigational site 34, Yamagata
  - Investigational site 04, Yamaguchi
  - Investigational site 26, Yamaguchi

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Continuous Infusion High-dose Group (Group H) | Continuous Infusion Low-dose Group (Group L) | Approved Dosing Regimen Group (Control Group)
Started | 7 | 4 | 6
Completed | 4 | 1 | 5
Not Completed | 3 | 3 | 1
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 0
Not completed — One subject of control group who discontinued prior to initiation of study drug administration. | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Among the randomised of 17 subjects, the baseline participants consisted of 15 subjects, excluding 1 who withdrew their consent after randomization and 1 who discontinued prior to initiation of study drug administration.
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Infusion High-dose Group (Group H) | Continuous Infusion Low-dose Group (Group L) | Approved Dosing Regimen Group (Control Group) | Total
Number analyzed (Participants) | 7 | 3 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.3 (6.8) | 75.7 (7.4) | 64.4 (11.2) | 72.2 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 3 | 11
  Male | 1 | 1 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 7 | 3 | 5 | 15
  Non-Japanese | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With National Institutes of Health Stroke Scale (NIHSS) Score Improved.
Description: NIHSS is a scale to objectively quantify the neurologic impairment caused by a stroke.
  Possible scores range from 0 (no stroke symptoms) to 40(severe stroke).
Time Frame: Baseline up to Day 7
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Infusion High-dose Group (Group H) | Continuous Infusion Low-dose Group (Group L) | Approved Dosing Regimen Group (Control Group)
Number analyzed (Participants) | 7 | 3 | 5
Participants
  Day 1 | 0 | 0 | 0
  Day 2 | 2 | 0 | 1
  Day 3 | 2 | 0 | 1
  Day 4 | 2 | 0 | 1
  Day 5 | 2 | 0 | 1
  Day 6 | 3 | 1 | 1
  Day 7 | 3 | 1 | 1

2. Secondary Outcome: Comparison of National Institutes of Health Stroke Scale (NIHSS)
Description: NIHSS is a scale used to objectively quantify the neurologic impairment caused by a stroke.
  Possible scores range from 0 (no stroke symptoms) to 40 (severe stroke).
Time Frame: Day 14, at discharge(from Day15 to after 3 months) and after 3 months
Population: Among the randomised of 17 subjects, the baseline participants consisted of 15 subjects, excluding 1 who withdrew their consent after randomization and 1 who discontinued prior to initiation of study drug administration. The number of participants decreased at each evaluation point because there was missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuous Infusion High-dose Group (Group H) | Continuous Infusion Low-dose Group (Group L) | Approved Dosing Regimen Group (Control Group)
Number analyzed (Participants) | 7 | 3 | 5
units on a scale
  Day 14: number analyzed (Participants) | 6 | 2 | 5
  Day 14 | 3.7 (6.1) | 2.5 (2.1) | 2.8 (1.5)
  at discharge: number analyzed (Participants) | 4 | 2 | 3
  at discharge | 3.5 (5.1) | 2.0 (1.4) | 3.3 (1.5)
  after 3 months: number analyzed (Participants) | 3 | 1 | 5
  after 3 months | 3.3 (3.2) | 0.0 (NA) — Standard Deviation not calculable for 1 participant. | 1.8 (0.8)

3. Secondary Outcome: Number of Participants With Modified Rankin Scale (mRS) 0-1 at Each Evaluations
Description: mRS is a scale for measuring the degree of disability caused by a stroke. Possible scores range from Grade 0 (no symptoms) to Grade 6 (death). Number of Participants with Modified Rankin Scale (mRS) 0-1 are evaluated.
Time Frame: at discharge(from Day15 to after 3 months) and after 3 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Infusion High-dose Group (Group H) | Continuous Infusion Low-dose Group (Group L) | Approved Dosing Regimen Group (Control Group)
Number analyzed (Participants) | 7 | 3 | 5
Participants
  at discharge: number analyzed (Participants) | 6 | 2 | 5
  at discharge | 4 | 1 | 3
  after 3 months: number analyzed (Participants) | 3 | 1 | 5
  after 3 months | 2 | 1 | 3

4. Secondary Outcome: Comparison of Barthel Index (BI)
Description: BI is a scale for measuring performance in Activities of Daily Living (ADL). Possible scores range from 0 (worst) to 100 (best).
Time Frame: at discharge(from Day15 to after 3 months) and after 3 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuous Infusion High-dose Group (Group H) | Continuous Infusion Low-dose Group (Group L) | Approved Dosing Regimen Group (Control Group)
Number analyzed (Participants) | 7 | 3 | 5
units on a scale
  at discharge: number analyzed (Participants) | 4 | 2 | 3
  at discharge | 80 (36.7) | 72.5 (38.9) | 83.3 (28.9)
  after 3 months: number analyzed (Participants) | 3 | 1 | 5
  after 3 months | 90 (17.3) | 100 (NA) — Standard Deviation not calculable for 1 participant. | 100 (0)

5. Secondary Outcome: Comparison of Functional Independence Measure (FIM)
Description: FIM is a scale used to evaluate the functional status. Possible scores range from 18 (worst) to 126 (best).
Time Frame: at discharge(from Day15 to after 3 months) and after 3 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuous Infusion High-dose Group (Group H) | Continuous Infusion Low-dose Group (Group L) | Approved Dosing Regimen Group (Control Group)
Number analyzed (Participants) | 7 | 3 | 5
units on a scale
  at discharge: number analyzed (Participants) | 6 | 2 | 5
  at discharge | 102.2 (33.8) | 91.5 (41.7) | 121.8 (4.1)
  after 3 months: number analyzed (Participants) | 3 | 1 | 5
  after 3 months | 93.7 (54.3) | 125.0 (NA) — Standard Deviation not calculable for 1 participant. | 123.4 (2.5)

ADVERSE EVENTS:
Time Frame: Adverse events occurring in subjects up to 3 months after the start of investigational product treatment were investigated.
Arm/Group | Continuous Infusion High-dose Group (Group H) | Continuous Infusion Low-dose Group (Group L) | Approved Dosing Regimen Group (Control Group)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/7 | 1/3 | 1/5
Other Adverse Events (participants affected / at risk) | 6/7 | 2/3 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Continuous Infusion High-dose Group (Group H) (N=7) | Continuous Infusion Low-dose Group (Group L) (N=3) | Approved Dosing Regimen Group (Control Group) (N=5)
Hepatic mass (Hepatobiliary disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Continuous Infusion High-dose Group (Group H) (N=7) | Continuous Infusion Low-dose Group (Group L) (N=3) | Approved Dosing Regimen Group (Control Group) (N=5)
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Dementia (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT03346538/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT03346538/SAP_001.pdf